CLINICAL TRIAL: NCT00404742
Title: A Double-Masked, Placebo-Controlled, Multi-Center, Parallel-Group, Dose-Ranging Study With an Optional Extension to Assess the Efficacy and Safety of LX211 as Therapy in Subjects With Clinically Quiescent Sight Threatening, Non-infectious Intermediate, Anterior and Intermediate, Posterior or Pan-Uveitis
Brief Title: A Study of LX211 in Clinically Quiescent Non-infectious Intermediate, Anterior and Intermediate, Posterior or Pan-Uveitis
Acronym: LUMINATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lux Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX211-02-UV; EudraCT No: 2006-006544-66
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Uveitis, Posterior; Uveitis, Intermediate; Panuveitis
Keywords: uveitis; calcineurin
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate; Panuveitis; Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- LX211, 0.2 mg/kg (Active Comparator)
  Interventions: Drug: LX211
- LX211, 0.4 mg/kg (Active Comparator)
  Interventions: Drug: LX211
- LX211, 0.6 mg/kg (Active Comparator)
  Interventions: Drug: LX211

INTERVENTIONS:
Drug: Placebo — PO BID
  Arms: Placebo
Drug: LX211 — 0.2 mg/kg, twice a day (BID)
  Arms: LX211, 0.2 mg/kg
Drug: LX211 — 0.4 mg/kg, twice a day (BID)
  Arms: LX211, 0.4 mg/kg
Drug: LX211 — 0.6 mg/kg, twice a day (BID)
  Arms: LX211, 0.6 mg/kg

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of LX211 as therapy in subjects with clinically quiescent non-infectious uveitis

ELIGIBILITY:
Inclusion Criteria:

* A documented history of non-infectious intermediate, anterior and intermediate, posterior or panuveitis.
* Minimum prescribed therapy upon enrollment is one or more of the following:

  * systemic prednisone or equivalent averaging ≥ 10 mg/day
  * at least 2 periocular/intravitreal corticosteroid administrations for control of inflammatory disease within the previous 8 months (but not within 6 weeks of randomization).
  * at least one, but not more than 2 immunosuppressive drugs from among the following compounds: cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, methotrexate
* Subjects with clinically quiescent uveitis in both eyes at enrollment and who have been on a stable treatment regimen for a minimum of 6 weeks
* Best-corrected distance visual acuity in the worst involved eye of 20/400 or better (ETDRS logMAR <1.34)
* Subjects not planning to undergo elective ocular surgery during the study

Exclusion Criteria:

* Evidence of active, uncontrolled non-infectious uveitis
* Periocular administration of corticosteroids within the previous 6 weeks.
* Uveitis of infectious etiology
* Uncontrolled glaucoma
* Clinically suspected or confirmed central nervous system or ocular lymphoma
* History or diagnosis of Behçet's disease
* Primary diagnosis of anterior uveitis

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
recurrence of ocular inflammation | 26 weeks

SECONDARY OUTCOMES:
BCVA | 26 weeks
systemic corticosteroid usage | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Anglade, M.D., Study Chair — Chief Medical Officer
Locations (41):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - University of Illinois - Chicago, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wilmer Eye Institute, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Massachusetts Eye Research and Surgery Institute, Cambridge, Massachusetts
  - Associated Retinal Consultants, PC, Grand Rapids, Michigan
  - Tauber Eye Center, Kansas City, Missouri
  - UMDNJ-New Jersey Medical School, Ophthalmology Dept., Newark, New Jersey
  - New York Eye & Ear Hospital, New York, New York
  - Duke University Eye Center, Erwin Road, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - Texas Retina Associates, Arlington, Texas
  - Brian B. Berger, MD, P.A., Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Retina & Uveitis Consultants of Texas, San Antonio, Texas
  - Viginia Eye Consultants, Norfolk, Virginia
- Austria (2):
  - Universitätsklinik für Augenheilkunde, Salzburg
  - Klinik für Augenheilkunde, Dept. of Ophthalmology, Vienna
- Canada (3):
  - Ivey Eye Institute, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec
- France (2):
  - Center Hospitalier Universitaire d' Angers, Service d'Opthalmologie, Angers
  - Hôpital Pitié Salpétrière, Service d'Ophtalmologie, Paris
- Germany (3):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Augenklinik der Universität Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
- India (9):
  - L V Prasad Eye Institute, Hyderabaad, Andhra Pradesh
  - Consultant, Retina and Vitreous Services, Bhubaneswar L V Prasad Eye Institute, Bhubaneswar, Odisha
  - Department of Opthalmology, Sankara Nethralaya, Medical Research Foundation,, Chennai, Tamil Nadu
  - Aravind Eye Hospitals and Postgraduate Institute of Ophthalmology, Madurai, Tamil Nadu
  - Vittala International Institute of Ophthalmology, Bangalore
  - Advanced Eye Centre, Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Aravind Eye Hospital, Uvea Clinic, Coimbatore
  - Aditya Jyot Eye Hospital Pvt Ltd, Mumbai
  - Dr. R. P. Centre for Ophthalmic Sciences, All India Institute of Medical Sciences, New Delhi
- United Kingdom (3):
  - Bristol Eye Hospital and University of Bristol, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital, London

REFERENCES:
- See also: Related Info — http://www.luxbio.com